CLINICAL TRIAL: NCT00369265
Title: A Randomized, Placebo-Controlled Assessment of Lansoprazole 30 mg Bid in the Treatment of Gastroesophageal Reflux Associated With Laryngitis
Brief Title: Safety and Efficacy of Lansoprazole 30mg Twice Daily in Treatment of Laryngitis Associated With Gastroesophageal Reflux
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Pharmaceutical company purchased by another company and funding was terminated.
Sponsor: American Institute for Voice and Ear Research (Other)
Responsible Party: Principal Investigator, Robert T. Sataloff, MD, M.D., D.M.A., FACS, American Institute for Voice and Ear Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10166
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Laryngopharyngeal Reflux
Keywords: Gastroesophageal reflux; Laryngitis; Hoarseness; Dysphonia; Proton pump inhibitor
MeSH Terms: conditions — Laryngopharyngeal Reflux; Gastroesophageal Reflux; Laryngitis; Hoarseness; Dysphonia | interventions — Lansoprazole; Sugars

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lansoprazole (Experimental): Lansoprazole 30 mg Twice Daily
  Interventions: Drug: Lansoprazole
- Sugar pill (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Sugar pill

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 30mg twice daily
  Arms: Lansoprazole
Dietary Supplement: Sugar pill — placebo twice daily
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether Lansoprazole 30mg taken twice daily is effective in the treatment of laryngitis due to gastroesophageal reflux.

DETAILED DESCRIPTION:
The investigators propose to study the effect of Lansoprazole 30 mg bid therapy vs. placebo in patients who present with symptoms characteristic of reflux laryngitis. The efficacy of Lansoprazole 30 mg bid in healing and improving reflux laryngitis will be determined. For the purpose of this study, healed reflux laryngitis will be defined as an improvement or resolution of arytenoid erythema and improvement in symptoms. Improved reflux laryngitis will be defined as improvement in any two of the following areas: arytenoid erythema; voice quality as assessed by the patients or health care provider; or, improvement/resolution of related symptoms (throat clearing, cough, etc.). The impact of Lansoprazole 30 mg bid therapy on quality of life will be evaluated in a preliminary fashion.

ELIGIBILITY:
Inclusion Criteria:

* Vocal skills necessary to complete test procedures reliably.
* Voice complaints and/or other symptoms suggestive of reflux laryngitis
* Signed informed consent
* At least 18 years of age.
* Complete medical history and physical examination within 30 days prior to initiation of the study drug.
* Laryngoscopy documenting laryngeal pathology compatible with moderate to severe reflux laryngitis (> grade 3 arytenoid erythema) within 30 days of initiation of the study drug.
* Gastroesophageal reflux confirmed by 24-hour (a minimum of 16 hours required for inclusion) pH impedance monitor.
* Ambulatory outpatient status.
* If female, a negative pregnancy test at the screening visit or either: i) surgically sterilized (bilateral tubal ligation or hysterectomy), or ii) at least 1 year post-menopausal, or iii) using acceptable methods of contraception in the presence of childbearing potential.

Exclusion Criteria:

* Concurrent laryngeal disease, if such disease or its treatment would interfere with evaluation of study results. For example, patients with mass lesions such as laryngeal cysts or laryngeal carcinoma will be excluded. Patients with acute laryngeal infections or acute laryngeal allergies will be excluded until these conditions have been resolved; but they may be considered for inclusion thereafter.
* Any upper gastroenterological or esophageal surgery except simple over-sewing of a perforated ulcer.
* Active substance abuse.
* Tobacco use.
* Known hypersensitivity or allergy to any protein pump inhibitor.
* ALT (SGPT) or AST (SGOT) greater than 2 times the upper limit of normal.
* Renal impairment (serum creatinine > 2.0 mg/dl).
* Any clinically significant, unstable medical condition.
* Use of any proton pump inhibitor within 7 days prior to 24-hour pH impedance monitoring or baseline strobovideolaryngoscopy, or use of H2 receptor antagonist during the 48 hours prior to 24-hour pH impedance monitoring or baseline strobovideolaryngoscopy.
* Use of an investigational drug or participation in an investigational study, within 30 days prior to starting study drug.
* Previous participation in this study.
* Pregnant women.
* Women breast feeding infants.
* Inability or refusal to follow directions.
* Open label sub-study has same inclusion and exclusion criteria, with exception that subjects should have: 1) Clinical diagnosis of non-acid reflux, with less than 5 episodes of proximal acid reflux, and 2) Symptoms and signs consistent with gastroesophageal reflux.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Sataloff, MD, DMA, Principal Investigator — American Institute for Voice and Ear Research
Locations (3):
- United States (3):
  - Henry Ford Hospital, Department of Otolaryngology, Detroit, Michigan
  - American Institute for Voice and Ear Research, Philadelphia, Pennsylvania
  - Cornell University, Van Lawrence Voice Center, Houston, Texas

REFERENCES:
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Belafsky PC, Postma GN, Koufman JA. Laryngopharyngeal reflux symptoms improve before changes in physical findings. Laryngoscope. 2001 Jun;111(6):979-81. doi: 10.1097/00005537-200106000-00009. PMID 11404607
- [Background] Bogdasarian RS, Olson NR. Posterior glottic laryngeal stenosis. Otolaryngol Head Neck Surg (1979). 1980 Nov-Dec;88(6):765-72. doi: 10.1177/019459988008800625. No abstract available. PMID 7208045
- [Background] Cherry J, Margulies SI. Contact ulcer of the larynx. Laryngoscope. 1968 Nov;78(11):1937-40. doi: 10.1288/00005537-196811000-00007. No abstract available. PMID 5722896
- [Background] Delahunty JE, Cherry J. Experimentally produced vocal cord granulomas. Laryngoscope. 1968 Nov;78(11):1941-7. doi: 10.1288/00005537-196811000-00008. No abstract available. PMID 5722897
- [Background] Eherer AJ, Habermann W, Hammer HF, Kiesler K, Friedrich G, Krejs GJ. Effect of pantoprazole on the course of reflux-associated laryngitis: a placebo-controlled double-blind crossover study. Scand J Gastroenterol. 2003 May;38(5):462-7. doi: 10.1080/00365520310001860. PMID 12795454
- [Background] El-Serag HB, Lee P, Buchner A, Inadomi JM, Gavin M, McCarthy DM. Lansoprazole treatment of patients with chronic idiopathic laryngitis: a placebo-controlled trial. Am J Gastroenterol. 2001 Apr;96(4):979-83. doi: 10.1111/j.1572-0241.2001.03681.x. PMID 11316215
- [Background] Koufman J, Sataloff RT, Toohill R. Laryngopharyngeal reflux: consensus conference report. J Voice. 1996 Sep;10(3):215-6. doi: 10.1016/s0892-1997(96)80001-4. No abstract available. PMID 8865091
- [Background] Morrison MD. Is chronic gastroesophageal reflux a causative factor in glottic carcinoma? Otolaryngol Head Neck Surg. 1988 Oct;99(4):370-3. doi: 10.1177/019459988809900403. PMID 3148885
- [Background] Noordzij JP, Khidr A, Evans BA, Desper E, Mittal RK, Reibel JF, Levine PA. Evaluation of omeprazole in the treatment of reflux laryngitis: a prospective, placebo-controlled, randomized, double-blind study. Laryngoscope. 2001 Dec;111(12):2147-51. doi: 10.1097/00005537-200112000-00013. PMID 11802014
- [Background] Vaezi MF, Richter JE, Stasney CR, Spiegel JR, Iannuzzi RA, Crawley JA, Hwang C, Sostek MB, Shaker R. Treatment of chronic posterior laryngitis with esomeprazole. Laryngoscope. 2006 Feb;116(2):254-60. doi: 10.1097/01.mlg.0000192173.00498.ba. PMID 16467715
- [Background] Wetmore RF. Effects of acid on the larynx of the maturing rabbit and their possible significance to the sudden infant death syndrome. Laryngoscope. 1993 Nov;103(11 Pt 1):1242-54. doi: 10.1288/00005537-199311000-00006. PMID 8231577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inadequate recruitment during this study; therefore, the study was terminated.
Groups:
- Sugar Pill: Placebo for Lansoprazole twice daily
Period: Overall Study
Arm/Group | Sugar Pill | Lansoprazole
Started | 4 | 7
Completed | 0 | 0
Not Completed | 4 | 7
Not completed — Study terminated | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Lansoprazole | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 33.0 (11.56) | 40.1 (17.33) | 37.5 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement or Resolution of Arytenoid Erythema
Description: Improvement was measured by score on an arytenoid erythema grading scale assigned by member of research staff and independent observers at 6 weeks
Time Frame: 6 weeks
Population: No results to report; Study was terminated
Arm/Group | Sugar Pill | Lansoprazole
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Lansoprazole
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7

LIMITATIONS AND CAVEATS:
The study was terminated due to inadequate subject recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No